CLINICAL TRIAL: NCT00618267
Title: Single Center, Pilot Study to Measure ATP Expression in Lymphocytes of MS Patients Undergoing Various Therapies by Means of Using the "ImmuKnow®" Test
Brief Title: ATP Expression in Lymphocytes of MS Patients by Means of "ImmuKnow®" Assay.
Acronym: Cylex
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Biogen Idec, Inc., Biogen Idec, Inc.
Other Study IDs: 014-07-NAT; Biogen Idec 014-07-NAT
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — About 1 ½ teaspoons of blood will be drawn.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to see if we can find a new way to test how certain Multiple Sclerosis (MS) medications work in the body and to better understand how the medicines change certain substances (cells) found in the immune (protective) system.

Blood test will be drawn by doing the following:

* Use a new method called the "Immuknow®" Test to see if this method will help to better understand how MS medicines work.
* Measure certain levels of immune cells in a new way, to see if it this will help to understand the body's response to MS medicines.

These methods will test those with MS who are not taking any MS medications, to help us compare the results.

About 100 subjects will be enrolled in this study at the Partners Multiple Sclerosis Center at Brigham and Women's Hospital. Biogen Idec, Inc. of Cambridge, MA, is paying for this study to be done.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effects of various therapies (immunomodulatory as well as immunosuppressive) on ATP levels in CD4+ cells and to determine whether the "ImmuKnow®" assay is an appropriate screening tool to assess the immunocompetence of potential Tysabri patients.

Secondary objective is to correlate the expression of ATP in CD4+ cells with CD4+ cell count.

Tertiary objective is to examine the level of regulatory T-cells (CD4+ and CD25+) in MS patients and its possible correlation to the therapy used, and how well a recently proposed marker of regulatory T-cells, LAP, correlates with CD25 marker.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be taking 1 of the following medications for 3 months or more: Cytoxan, Cellcept, Novantrone Betaseron, Rebif, Avonex or Copaxone.
2. Patients must be able to provide written informed consent.

Exclusion Criteria:

1. Patients on combination of multiple medications.
2. Restricted treatment whereby no use in 50 days prior to enrollment visit is permitted: systemic steroids.
3. With educational completion below 8th grade school equivalent or non-fluent in English.
4. Any other reason, in the opinion of both the Investigator and/or Sponsor, the patient is determined not suitable for study participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Multiple Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the effects of various therapies (immunomodulatory as well as immunosuppressive) on ATP levels in CD4+ cells. | 1 blood draw

SECONDARY OUTCOMES:
Secondary objective is to correlate the expression of ATP in CD4+ cells with CD4+ cell count. | 1 blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Samia J Khoury, MD, Principal Investigator — Harvard Medical School, Brigham and Women's Hospital - Partners MS Center
Locations (1):
- Brigham and Women's Hospital - Partners MS Center, Brookline, Massachusetts, United States